CLINICAL TRIAL: NCT03098303
Title: Criteria Associated With Patient Willingness to Participate in Biomedical Research: a Prospective, Observational Study
Brief Title: Criteria Associated With Patient Willingness to Participate in Biomedical Research
Acronym: PROTOACCEPT
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9373; 2014-A01201-46 (Other: RCB number)
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Consulting in Pneumology Department, But Not for Oncology or Tobacology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to determine the variables associated with patient acceptation or refusal to participate in a clinical research protocol when seen in during a pneumology consultation (excluding oncology and tobaccology).

DETAILED DESCRIPTION:
The secondary objectives of this study are:

* To compare patient acceptance rates for participation in a clinical research protocol before and after January 15, 2016.
* To determine the variables associated with accepting or refusing to participate in a clinical research protocol for patients seen during a pneumology consultation (excluding oncology and tobaccology) before January 15, 2016.
* To determine the variables associated with accepting or refusing to participate in a clinical research protocol for patients seen during a pneumology consultation (excluding oncology and tobaccology) after January 15, 2016.
* To describe the patient population seen during pneumology consultations.
* To determine the variables associated with accepting or refusing to participate in a clinical research protocol sponsored by a pharmaceutical laboratory.
* To determine the variables associated with accepting or refusing to participate in a clinical research protocol sponsored by an academic institution.
* Construct clusters (homogeneous groups) of patients seen during the pneumology consultations.

ELIGIBILITY:
Inclusion Criteria:

* The patient was informed about the study.
* The patient is scheduled for a consult in the pneumology department

Exclusion Criteria:

* The patient is under judicial protection or is an adult under any kind of guardianship
* The patient expresses opposition to the study
* It is impossible to correctly inform the patient about the study
* The patient cannot fluently read French
* The patient is pregnant
* The patient is breastfeeding
* The patient has cancer
* The patient is consulting in tabaccology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population corresponds to patients with respiratory disease. This study will be proposed to all patients consulting (excluding oncology and tobacco) in the associated departments.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-12-23 (Actual); Primary Completion 2016-12-13 (Actual); Study Completion 2016-12-13 (Actual)

PRIMARY OUTCOMES:
Acceptation or refusal to participate in a biomedical research study | Day 0 (cross-sectional study)
  Positive or negative response to the question "If a biomedical research protocole were proposed to you, would you accept to participate?"

SECONDARY OUTCOMES:
The PROTOACCEPT questionnaire | Day 0 (cross-sectional study)
  The PROTOACCEPT questionnaire (see links below).

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bourdin, MD, PhD, Study Director — Montpellier University Hospitals
Locations (4):
- France (4):
  - Polyclinique Saint-Privat, Boujan-sur-Libron
  - Clinique de Marignane, Marignane
  - APHM - Hôpital Nord, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier

REFERENCES:
- [Result] Pahus L, Suehs CM, Halimi L, Bourdin A, Chanez P, Jaffuel D, Marciano J, Gamez AS, Vachier I, Molinari N. Patient distrust in pharmaceutical companies: an explanation for women under-representation in respiratory clinical trials? BMC Med Ethics. 2020 Aug 13;21(1):72. doi: 10.1186/s12910-020-00509-y. PMID 32791969
- [Result] Molinari N, Suehs C, Vachier I, Pahus L, Halimi L, Gamez AS, Chanez P, Bourdin A. Adverse publicity of serious side effects to healthy volunteers has limited effect on willingness-to-participate in clinical trials. Clin Trials. 2019 Aug;16(4):440-442. doi: 10.1177/1740774519840268. Epub 2019 Mar 29. No abstract available. PMID 30922104
- See also: The PROTOACCEPT patient questionnaire — https://osf.io/gccjd/
- See also: PROTOACCEPT on the Open Science Framework — https://osf.io/nsjjr/